CLINICAL TRIAL: NCT03164564
Title: A Phase 3 Double Blind Safety and Efficacy Study of Long-Acting Injectable Cabotegravir Compared to Daily Oral TDF/FTC for Pre-Exposure Prophylaxis in HIV-Uninfected Women
Brief Title: Evaluating the Safety and Efficacy of Long-Acting Injectable Cabotegravir Compared to Daily Oral TDF/FTC for Pre-Exposure Prophylaxis in HIV-Uninfected Women
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HPTN 084; 38070 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Results first posted 2023-03-28 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — cabotegravir; Tenofovir; Emtricitabine; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: CAB + Placebo TDF/FTC + CAB LA (Experimental): During Step 1, participants will receive daily oral CAB and oral TDF/FTC placebo for 5 weeks. In Step 2, participants will receive injections of CAB LA at two time points 4 weeks apart and every 8 weeks thereafter and daily oral TDF/FTC placebo beginning at Week 5. In Step 3, participants will receive daily TDF/FTC for up to 48 weeks, starting no later than 8 weeks after the last injection.
  Interventions: Drug: Oral CAB; Drug: Oral TDF/FTC; Drug: Placebo for oral TDF/FTC; Drug: CAB LA
- Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA (Active Comparator): During Step 1, participants will receive daily TDF/FTC and oral CAB placebo for 5 weeks. In Step 2, participants will receive daily TDF/FTC and placebo for CAB LA injections at two times points 4 weeks apart and every 8 weeks thereafter beginning at Week 5. In Step 3, participants will receive daily TDF/FTC for up to 48 weeks, starting no later than 8 weeks after the last injection.
  Interventions: Drug: Oral TDF/FTC; Drug: Placebo for oral CAB; Drug: Placebo for CAB LA

INTERVENTIONS:
Drug: Oral CAB — CAB 30 mg tablet
  Other Names: Cabotegravir
  Arms: Arm A: CAB + Placebo TDF/FTC + CAB LA
Drug: Oral TDF/FTC — TDF/FTC 300 mg/200 mg fixed dose combination tablet
  Other Names: Tenofovir disoproxil fumarate/emtricitabine; Truvada
Drug: Placebo for oral CAB — Placebo tablets
  Arms: Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA
Drug: Placebo for oral TDF/FTC — Placebo tablets
  Arms: Arm A: CAB + Placebo TDF/FTC + CAB LA
Drug: CAB LA — 600 mg administered as one 3 mL (600 mg) intramuscular injection in the gluteal muscle
  Other Names: Cabotegravir long-acting injectable
  Arms: Arm A: CAB + Placebo TDF/FTC + CAB LA
Drug: Placebo for CAB LA — Administered as one 3 mL intramuscular injection in the gluteal muscle
  Arms: Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA

SUMMARY:
This study will evaluate the safety and efficacy of the long-acting injectable agent cabotegravir (CAB LA) compared to daily oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) for pre-exposure prophylaxis (PrEP) in HIV-uninfected women.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of the long-acting injectable integrase inhibitor cabotegravir (CAB LA) compared to daily oral tenofovir disoproxil fumarate/emtricitabine (TDF/FTC) for pre-exposure prophylaxis (PrEP) in a population of sexually active HIV-uninfected women at risk for HIV.

This study will take place in three steps. Participants will be randomly assigned to one of two arms:

Arm A:

Step 1: Participants will receive daily oral CAB and TDF/FTC placebo for 5 weeks.

Step 2: Participants will receive injections of CAB LA at two time points 4 weeks apart and every 8 weeks thereafter and daily TDF/FTC placebo beginning at Week 5.

Arm B:

Step 1: Participants will receive daily TDF/FTC and oral CAB placebo for 5 weeks.

Step 2: Participants will receive daily TDF/FTC and intramuscular (IM) placebo injections at two time points 4 weeks apart and every 8 weeks thereafter beginning at Week 5.

Step 2 will continue until the last enrolled participant reaches approximately 76 weeks on Step 2 (Week 81 for the last enrolled participant).

In Step 3, all participants (Arms A and B) will receive daily TDF/FTC for up to 48 weeks, starting no later than 8 weeks after the last injection.

At the end of Step 3, all participants will then transition to locally available HIV prevention services, including services for PrEP, if available.

Study visits will occur at Day 0 and at Weeks 2 and 4 during Step 1. During Step 2, participants will attend up to 24 visits, depending on when they enroll in the study. Study visits will occur every 12 weeks during Step 3. Study visits may include physical examinations; blood, urine, and vaginal swab collection; risk reduction, adherence counseling, and contraception counseling.

HPTN 084-01 is a sub-study of HPTN 084. The purpose of this study is to examine the safety, tolerability, and acceptability of CAB LA for the prevention of HIV among adolescent females. Participants will receive oral CAB for 5 weeks, followed by 34 weeks on CAB LA, then quarterly visits for 48 weeks after final injection. All participants who have received at least one injection will be followed for 48 weeks after their last injection. Total study duration per participant will be approximately 21 months.

ELIGIBILITY:
Inclusion Criteria:

* Born female
* 18-45 years at the time of screening
* Willing and able to provide informed consent
* Willing and able to undergo all required study procedures
* Non-reactive HIV test results at Screening and Enrollment. Note: HIV-uninfected, based on HIV test results obtained at Screening and just prior to randomization at the Enrollment visit. All HIV test results from the Screening visit must be obtained and must all be negative/non-reactive. This includes testing for acute HIV infection, which must be performed within 14 days of Enrollment. In addition, at least one HIV test result using blood drawn at the Enrollment visit must be obtained prior to randomization into the study and must be negative/non-reactive. Individuals who have one or more reactive or positive HIV test result(s) will not be enrolled, even if subsequent confirmatory testing indicates that they are not HIV-infected (see SSP Manual). Those with any enrollment HIV test result positive will proceed through the HIV algorithm per the SSP but will not be able to receive study product regardless of subsequent test results.
* Sexually active (i.e., vaginal intercourse on a minimum of two separate days in the 30 days prior to Screening)
* Score of greater than or equal to 5 using a modified VOICE risk score
* No plans to re-locate or travel away from the site for greater than or equal to 8 consecutive weeks during study participation
* Creatinine clearance of greater than or equal to 60 mL/min (using Cockcroft-Gault equation) (use sex at birth for calculation)

  * Although not protocol exclusionary, sites should carefully consider the advisability of enrolling participants with calculated creatinine clearance between 60-70 mL/min, as limited changes in creatinine clearance during study conduct will lead to protocol-mandated product holds and may alter the risk-benefit considerations of study participation
* Hepatitis B virus (HBV) surface antigen (HBsAg) negative and accepts vaccination
* Alanine aminotransferase (ALT) less than 2 x upper limit of normal (ULN) and total bilirubin (Tbili) less than or equal to 2.5 x ULN
* HCV antibody negative
* If of reproductive potential (defined as pre-menopausal women who have not had a sterilization procedure per self-report, such as hysterectomy, bilateral oophorectomy, tubal ligation or salpingectomy), must have a negative beta human chorionic gonadotropin (βHCG) pregnancy test (sensitivity of less than or equal to 25 mIU/mL) performed (and results known) on the same day as and before initiating the protocol-specified study product(s) at Enrollment.
* Have documented evidence of surgical sterilization, OR documented evidence of no uterus (e.g., hysterectomy), OR must agree to use a reliable form of long acting contraception, during the trial and for 52 weeks after stopping the long acting injectable, or 30 days after stopping oral study product, from the list below:

  * Intrauterine device (IUD) or intrauterine system (IUS) that meets less than 1% failure rate as stated in the product label
  * Hormone-based contraceptive that meets less than 1% failure rate when used consistently and correctly as stated in the product label (implants or injectables only; this excludes combined oral contraception)
* No medical condition that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records)
* No alcohol or substance use that, in the opinion of the study investigator, would interfere with the conduct of the study (e.g., provided by self-report, or found upon medical history and examination or in available medical records)

Exclusion Criteria:

* One or more reactive HIV test results at Screening or Enrollment, even if HIV infection is not confirmed
* Pregnant or currently breastfeeding, or intends to become pregnant and/or breastfeed during the study
* Co-enrollment in any other HIV interventional research study (provided by self-report or other available documentation), with one exception: IMPAACT 2026 (co-enrollment in IMPAACT 2026 is permitted for participants who become pregnant)
* Current or past enrollment in an HIV vaccine or broadly neutralizing antibody trial
* Current or chronic history of liver disease (e.g., non-alcoholic or alcoholic steatohepatitis) or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome, asymptomatic gallstones, or cholecystectomy)
* History of seizure disorder, per self-report
* Clinically significant cardiovascular disease, as defined by history/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PTCA) or any clinically significant cardiac disease
* Inflammatory skin conditions that compromise the safety of IM injections, per the discretion of the Investigator of Record (IoR). Mild skin conditions may not be exclusionary at the discretion of the IoR or designee
* Has a tattoo or other dermatological condition overlying the buttock region which in the opinion of the IoR or designee may interfere with interpretation of injection site reactions (ISRs)
* Coagulopathy (primary or iatrogenic) which would contraindicate IM injection
* Active or planned use of prohibited medications as described in the Investigator Brochure (IB) or listed in the Study Specific Procedures Manual (SSP) (provided by self-report, or obtained from medical history or medical records)
* Known or suspected allergy to study product components (active or placebo), including egg or soy products (egg and soy products are contained in Intralipid)
* If potentially able to conceive, unwilling to adhere to long acting contraception (IUD/IUS, injection, or implant) with a less than 1% failure rate when used consistently and correctly as stated in the product package insert/ manufacturer's guidelines

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3224 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2020-11-05 (Actual); Study Completion 2026-10-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sinead Delany-Moretlwe, PhD, DTM&H, Study Chair — Wits Reproductive Health and HIV Institute CRS (WRHI CRS); Mina Hosseinipour, MD, MPH, Study Chair — University of North Carolina (UNC) Project-Malawi, Tidziwe Centre
Locations (20):
- Gaborone CRS, Gaborone, South-East District, Botswana
- Eswatini Prevention Center CRS, Mbabane, Eswatini
- Kisumu Crs, Kisumu, Nyanza, Kenya
- Malawi (2):
  - Malawi CRS, Lilongwe, Central Region
  - Blantyre CRS, Blantyre
- South Africa (7):
  - Soweto HPTN CRS, Johannesburg, Gauteng
  - Ward 21 CRS, Johannesburg, Gauteng
  - Botha's Hill CRS, Durban, KwaZulu-Natal
  - Isipingo CRS, Isipingo, KwaZulu-Natal
  - Verulam CRS, Verulam, KwaZulu-Natal
  - Desmond Tutu TB Centre - Stellenbosch University (DTTC-SU) CRS, Cape Town, Western Cape
  - Emavundleni CRS, Cape Town, Western Cape
- Uganda (3):
  - UVRI-IAVI HIV Vaccine Program LTD. CRS, Entebbe
  - Baylor-Uganda CRS, Kampala
  - MU-JHU Research Collaboration (MUJHU CARE LTD) CRS, Kampala
- Zimbabwe (5):
  - Zengeza CRS, Chitungwiza, Mashonaland East Province
  - Seke South CRS, Chitungwiza
  - St Mary's CRS, Chitungwiza
  - Milton Park CRS, Harare
  - Spilhaus CRS, Harare

REFERENCES:
- [Derived] Marzinke MA, Han K, Hanscom B, Guo X, Piwowar-Manning E, Hendrix CW, Rose S, Spooner E, Mathew C, Innes S, Sekabira R, Mutambanengwe M, Rooney JF, Rinehart AR, Adeyeye A, Cohen MS, Hosseinipour M, Ford SL, Delany-Moretlwe S. Pharmacologic evaluation of delayed long-acting cabotegravir administration among cisgender women in HPTN 084. Antimicrob Agents Chemother. 2024 Nov 6;68(11):e0099424. doi: 10.1128/aac.00994-24. Epub 2024 Sep 23. PMID 39311597
- [Derived] Delany-Moretlwe S, Hughes JP, Bock P, Ouma SG, Hunidzarira P, Kalonji D, Kayange N, Makhema J, Mandima P, Mathew C, Spooner E, Mpendo J, Mukwekwerere P, Mgodi N, Ntege PN, Nair G, Nakabiito C, Nuwagaba-Biribonwoha H, Panchia R, Singh N, Siziba B, Farrior J, Rose S, Anderson PL, Eshleman SH, Marzinke MA, Hendrix CW, Beigel-Orme S, Hosek S, Tolley E, Sista N, Adeyeye A, Rooney JF, Rinehart A, Spreen WR, Smith K, Hanscom B, Cohen MS, Hosseinipour MC; HPTN 084 study group. Cabotegravir for the prevention of HIV-1 in women: results from HPTN 084, a phase 3, randomised clinical trial. Lancet. 2022 May 7;399(10337):1779-1789. doi: 10.1016/S0140-6736(22)00538-4. Epub 2022 Apr 1. PMID 35378077
- [Derived] Scarsi KK. Chasing the cabotegravir tail: implications for prevention. Lancet HIV. 2020 Jul;7(7):e451-e453. doi: 10.1016/S2352-3018(20)30165-X. Epub 2020 Jun 1. No abstract available. PMID 32497490

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: CAB + Placebo TDF/FTC + CAB LA | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA
Started | 1614 | 1610
Ongoing (Ongoing in the study indicates the participant has not terminated or completed the study.) | 1586 | 1586
Terminated From the Study (Excludes participants who completed the study.) | 25 | 17
Completed (Any seroconverters (per Site results or EAC) in Step 1 and seroconverters in Step 2 who have completed 48 weeks of follow-up.) | 3 | 7
Not Completed | 1611 | 1603
Not completed — Death | 3 | 0
Not completed — Withdrawal by Subject | 20 | 15
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Ongoing | 1586 | 1586

BASELINE CHARACTERISTICS:
Population: Overall enrolled participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: CAB + Placebo TDF/FTC + CAB LA | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA | Total
Number analyzed (Participants) | 1614 | 1610 | 3224
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25.0 [22.0 to 29.0] | 25.0 [22.0 to 30.0] | 25.0 [22.0 to 30.0]
Age, Customized [Count of Participants; unit: Participants]
  <25 | 800 | 794 | 1594
  >=25 | 814 | 816 | 1630
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1614 | 1610 | 3224
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1614 | 1610 | 3224
  Unknown or Not Reported | 0 | 0 | 0
Country [Count of Participants; unit: Participants]
  Botswana | 46 | 45 | 91
  Kenya | 31 | 35 | 66
  Malawi | 113 | 111 | 224
  South Africa | 653 | 655 | 1308
  Swaziland | 80 | 80 | 160
  Uganda | 300 | 296 | 596
  Zimbabwe | 391 | 388 | 779
Race [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Black or African American | 1612 | 1606 | 3218
  Mixed Race | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  White | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Pariicipants With Documented Incident HIV Infections
Description: The number of participants with an incident HIV infection that is confirmed by the HPTN Laboratory Center and Endpoint Adjudication Committee.
Time Frame: HIV tests at enrollment, weeks 2, 4, and 5, then every 4 weeks through week 25, then every 8 weeks. Analyzed through week 185 or the date of DSMB decision to unblind all participants, whichever is earliest.
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CAB + Placebo TDF/FTC + CAB LA | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA
Number analyzed (Participants) | 1614 | 1610
Participants | 4 | 36

2. Primary Outcome: Number of Participants Who Experienced Grade 2 or Higher Clinical and Laboratory Adverse Events (AEs) in Steps 1 and 2
Description: AEs will be summarized using MedDRA System Organ Class and preferred terms.
Time Frame: Treatment emergent AE measured with onset date through participant's last study visit, or the date of DSMB decision to unblind all participants, whichever is earliest. Assessed at each visit (injections visits q 8 weeks and safety visits q 8 weeks)
Population: All enrolled participants
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: CAB + Placebo TDF/FTC + CAB LA | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA
Number analyzed (Participants) | 1614 | 1610
Participants | 1487 | 1486

ADVERSE EVENTS:
Time Frame: Treatment emergent AE measured with onset date through participant's last study visit (up to 48 weeks after the last injection visit), or the date of DSMB decision to unblind all participants, whichever is earliest. Assessed at each visit (injections visits q 8 weeks and safety visits q 8 weeks)
Description: Adverse events are not reported separately for Step 1 (oral lead-in), Step 2 (CAB-LA injections or oral TDF/FTC) and Step 3 (open-label TDF/FTC) as an AE may not be reliably attributed to a specific step in the sequence.
Arm/Group | Arm A: CAB + Placebo TDF/FTC + CAB LA | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA
All-Cause Mortality (participants affected / at risk) | 3/1614 | 0/1610
Serious Adverse Events (participants affected / at risk) | 33/1614 | 33/1610
Other Adverse Events (participants affected / at risk) | 1486/1614 | 1486/1610
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: CAB + Placebo TDF/FTC + CAB LA (N=1614) | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA (N=1610)
Any Event in SOC (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Any Event in SOC (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Any Event in SOC (Gastrointestinal disorders) | 0 (0) | 2 (2)
Peptic ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Any Event in SOC (Hepatobiliary disorders) | 1 (1) | 2 (2)
Hepatitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (1)
Any Event in SOC (Infections and infestations) | 12 (13) | 11 (12)
Appendiceal abscess (Infections and infestations) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Endometritis (Infections and infestations) | 1 (1) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Gastritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis A (Infections and infestations) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 5 (5) | 3 (3)
Pelvic inflammatory disease (Infections and infestations) | 1 (1) | 2 (2)
Peritonsillar abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Tonsillitis bacterial (Infections and infestations) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Any Event in SOC (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Intentional overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Any Event in SOC (Investigations) | 1 (1) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 2 (2)
Any Event in SOC (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Any Event in SOC (Nervous system disorders) | 2 (3) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (2) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 8 (8) | 1 (1)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Preterm premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Ruptured ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Any Event in SOC (Psychiatric disorders) | 3 (4) | 5 (8)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Intentional self-injury (Psychiatric disorders) | 1 (1) | 1 (2)
Major depression (Psychiatric disorders) | 0 (0) | 1 (1)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Any Event in SOC (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: CAB + Placebo TDF/FTC + CAB LA (N=1614) | Arm B: TDF/FTC + Placebo CAB + Placebo CAB LA (N=1610)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 5 (5)
Any Event in SOC (Blood and lymphatic system disorders) | 40 (54) | 27 (28)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 4 (7) | 3 (4)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 2 (3) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (3) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Microcytic anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 22 (26) | 9 (9)
Thrombocytopenia (Blood and lymphatic system disorders) | 5 (5) | 3 (3)
Any Event in SOC (Cardiac disorders) | 1 (1) | 4 (4)
Palpitations (Cardiac disorders) | 0 (0) | 3 (3)
Rheumatic heart disease (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Any Event in SOC (Ear and labyrinth disorders) | 9 (9) | 5 (5)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 5 (5) | 2 (2)
Ear pruritus (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eustachian tube obstruction (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Otorrhoea (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Any Event in SOC (Endocrine disorders) | 1 (1) | 1 (1)
Goitre (Endocrine disorders) | 1 (1) | 1 (1)
Any Event in SOC (Eye disorders) | 47 (59) | 38 (42)
Asthenopia (Eye disorders) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 1 (1) | 0 (0)
Blindness unilateral (Eye disorders) | 0 (0) | 1 (1)
Chalazion (Eye disorders) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 31 (40) | 23 (26)
Dry eye (Eye disorders) | 4 (4) | 1 (1)
Eye allergy (Eye disorders) | 2 (2) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 1 (1)
Eye pruritus (Eye disorders) | 3 (3) | 5 (5)
Eyelid cyst (Eye disorders) | 0 (0) | 1 (1)
Periorbital swelling (Eye disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 2 (2) | 0 (0)
Pingueculitis (Eye disorders) | 0 (0) | 1 (1)
Refraction disorder (Eye disorders) | 1 (1) | 0 (0)
Scleritis allergic (Eye disorders) | 2 (2) | 2 (2)
Vernal keratoconjunctivitis (Eye disorders) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 4 (4) | 4 (4)
Abdominal pain (Gastrointestinal disorders) | 41 (42) | 41 (45)
Abdominal pain lower (Gastrointestinal disorders) | 19 (19) | 23 (23)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 11 (11)
Abdominal tenderness (Gastrointestinal disorders) | 0 (0) | 2 (2)
Acute abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 2 (2) | 2 (2)
Anal pruritus (Gastrointestinal disorders) | 0 (0) | 1 (1)
Any Event in SOC (Gastrointestinal disorders) | 334 (487) | 369 (574)
Aphthous ulcer (Gastrointestinal disorders) | 2 (3) | 0 (0)
Breath odour (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 18 (19) | 22 (25)
Dental caries (Gastrointestinal disorders) | 34 (36) | 51 (52)
Diarrhoea (Gastrointestinal disorders) | 56 (61) | 53 (56)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 (2) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 61 (82) | 71 (80)
Enteritis (Gastrointestinal disorders) | 6 (7) | 13 (13)
Food poisoning (Gastrointestinal disorders) | 10 (10) | 7 (7)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 67 (77) | 66 (79)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 (22) | 20 (27)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 12 (14) | 7 (7)
Hyperchlorhydria (Gastrointestinal disorders) | 8 (9) | 11 (17)
Lip blister (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 2 (2) | 3 (3)
Nausea (Gastrointestinal disorders) | 18 (19) | 41 (45)
Peptic ulcer (Gastrointestinal disorders) | 7 (7) | 8 (9)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 2 (2)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tooth impacted (Gastrointestinal disorders) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 21 (24) | 25 (25)
Vomiting (Gastrointestinal disorders) | 11 (12) | 29 (30)
Any Event in SOC (General disorders) | 75 (85) | 94 (102)
Chills (General disorders) | 2 (2) | 4 (4)
Complication of device removal (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 14 (15) | 13 (14)
Implant site induration (General disorders) | 0 (0) | 1 (1)
Implant site pain (General disorders) | 2 (2) | 4 (4)
Influenza like illness (General disorders) | 37 (40) | 44 (47)
Malaise (General disorders) | 3 (3) | 4 (5)
Medical device pain (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 5 (6) | 5 (5)
Peripheral swelling (General disorders) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 7 (8) | 10 (11)
Suprapubic pain (General disorders) | 0 (0) | 1 (1)
Swelling (General disorders) | 0 (0) | 2 (2)
Swelling face (General disorders) | 0 (0) | 1 (1)
Vessel puncture site pain (General disorders) | 3 (3) | 1 (1)
Any Event in SOC (Hepatobiliary disorders) | 2 (3) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 (3) | 1 (1)
Liver disorder (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergy to arthropod bite (Immune system disorders) | 1 (1) | 0 (0)
Any Event in SOC (Immune system disorders) | 34 (40) | 37 (48)
Atopy (Immune system disorders) | 0 (0) | 2 (2)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 1 (1) | 2 (2)
Hypersensitivity (Immune system disorders) | 6 (6) | 8 (8)
Multiple allergies (Immune system disorders) | 1 (1) | 2 (3)
Seasonal allergy (Immune system disorders) | 25 (31) | 26 (32)
Abdominal infection (Infections and infestations) | 1 (1) | 1 (2)
Abortion infected (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 2 (2) | 5 (5)
Abscess bacterial (Infections and infestations) | 1 (1) | 2 (2)
Abscess limb (Infections and infestations) | 0 (0) | 9 (9)
Abscess neck (Infections and infestations) | 1 (1) | 0 (0)
Abscess oral (Infections and infestations) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 16 (18) | 10 (10)
Acne pustular (Infections and infestations) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 5 (6) | 0 (0)
Amoebiasis (Infections and infestations) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Any Event in SOC (Infections and infestations) | 985 (2797) | 987 (2775)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 5 (5) | 0 (0)
Bacterial abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Bacterial blepharitis (Infections and infestations) | 1 (1) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 4 (4) | 1 (1)
Bacterial rhinitis (Infections and infestations) | 1 (1) | 1 (1)
Bacterial vaginosis (Infections and infestations) | 38 (43) | 36 (41)
Bacteriuria (Infections and infestations) | 0 (0) | 1 (1)
Bartholin's abscess (Infections and infestations) | 2 (2) | 2 (2)
Bartholinitis (Infections and infestations) | 0 (0) | 2 (2)
Body tinea (Infections and infestations) | 44 (56) | 34 (43)
Bronchitis (Infections and infestations) | 2 (2) | 4 (5)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1)
Burn infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1)
Candida infection (Infections and infestations) | 1 (1) | 3 (3)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 10 (10) | 6 (6)
Cervicitis (Infections and infestations) | 4 (4) | 3 (3)
Chancroid (Infections and infestations) | 1 (1) | 0 (0)
Chlamydial infection (Infections and infestations) | 115 (126) | 141 (159)
Chronic sinusitis (Infections and infestations) | 1 (1) | 0 (0)
Conjunctivitis (Infections and infestations) | 27 (33) | 29 (35)
Conjunctivitis bacterial (Infections and infestations) | 3 (3) | 6 (6)
Cystitis (Infections and infestations) | 7 (7) | 6 (6)
Cystitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Dermatitis infected (Infections and infestations) | 2 (2) | 1 (1)
Dermatophytosis (Infections and infestations) | 0 (0) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 4 (5) | 4 (4)
Dysentery (Infections and infestations) | 3 (3) | 1 (1)
Ear infection (Infections and infestations) | 0 (0) | 3 (3)
Ear infection fungal (Infections and infestations) | 2 (2) | 0 (0)
Endometritis (Infections and infestations) | 2 (2) | 2 (2)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Eye abscess (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 2 (2)
Eyelid infection (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 8 (8) | 7 (7)
Folliculitis (Infections and infestations) | 19 (20) | 14 (15)
Fungal infection (Infections and infestations) | 2 (2) | 0 (0)
Fungal skin infection (Infections and infestations) | 31 (33) | 26 (28)
Furuncle (Infections and infestations) | 2 (2) | 3 (3)
Gastric infection (Infections and infestations) | 1 (1) | 0 (0)
Gastritis bacterial (Infections and infestations) | 6 (6) | 7 (7)
Gastroenteritis (Infections and infestations) | 77 (97) | 74 (84)
Gastroenteritis bacterial (Infections and infestations) | 29 (35) | 28 (32)
Gastroenteritis shigella (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 2 (3) | 6 (6)
Genital abscess (Infections and infestations) | 0 (0) | 1 (1)
Genital candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Genital herpes (Infections and infestations) | 4 (4) | 7 (7)
Genital herpes simplex (Infections and infestations) | 1 (1) | 0 (0)
Genital infection (Infections and infestations) | 2 (2) | 1 (1)
Genital infection fungal (Infections and infestations) | 0 (0) | 1 (1)
Genital ulcer syndrome (Infections and infestations) | 0 (0) | 1 (1)
Genitourinary chlamydia infection (Infections and infestations) | 146 (169) | 151 (172)
Genitourinary tract gonococcal infection (Infections and infestations) | 67 (71) | 69 (77)
Genitourinary tract infection (Infections and infestations) | 5 (5) | 0 (0)
Gingivitis (Infections and infestations) | 3 (3) | 8 (8)
Gonococcal infection (Infections and infestations) | 39 (40) | 41 (43)
Gonorrhoea (Infections and infestations) | 20 (20) | 16 (17)
Groin abscess (Infections and infestations) | 0 (0) | 1 (1)
Helicobacter gastritis (Infections and infestations) | 2 (2) | 2 (2)
Helicobacter infection (Infections and infestations) | 1 (1) | 0 (0)
Helminthic infection (Infections and infestations) | 3 (3) | 2 (2)
Hepatitis A (Infections and infestations) | 0 (0) | 2 (2)
Hepatitis C (Infections and infestations) | 3 (3) | 2 (2)
Herpes simplex (Infections and infestations) | 1 (1) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 6 (6) | 2 (2)
Impetigo (Infections and infestations) | 3 (3) | 2 (2)
Implant site infection (Infections and infestations) | 0 (0) | 1 (1)
Infected cyst (Infections and infestations) | 2 (2) | 0 (0)
Infected skin ulcer (Infections and infestations) | 3 (3) | 0 (0)
Influenza (Infections and infestations) | 30 (31) | 22 (23)
Laryngitis (Infections and infestations) | 5 (5) | 0 (0)
Laryngitis viral (Infections and infestations) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 7 (7) | 11 (12)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 1 (1)
Lymphadenitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Malaria (Infections and infestations) | 50 (51) | 63 (79)
Mastitis (Infections and infestations) | 7 (7) | 5 (5)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1)
Mumps (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 75 (108) | 86 (133)
Nematodiasis (Infections and infestations) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 4 (4) | 2 (2)
Ophthalmic herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Oral bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Oral herpes (Infections and infestations) | 12 (13) | 10 (10)
Oral infection (Infections and infestations) | 0 (0) | 2 (2)
Oropharyngeal candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 2 (2) | 1 (1)
Otitis externa bacterial (Infections and infestations) | 0 (0) | 1 (1)
Otitis media (Infections and infestations) | 10 (10) | 8 (9)
Otitis media acute (Infections and infestations) | 5 (5) | 2 (3)
Otitis media bacterial (Infections and infestations) | 1 (1) | 2 (2)
Otitis media chronic (Infections and infestations) | 1 (1) | 0 (0)
Papilloma viral infection (Infections and infestations) | 2 (2) | 1 (2)
Parasitic gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 6 (6) | 3 (3)
Parotitis (Infections and infestations) | 1 (1) | 0 (0)
Pelvic infection (Infections and infestations) | 2 (2) | 2 (2)
Pelvic inflammatory disease (Infections and infestations) | 52 (58) | 44 (57)
Peptic ulcer helicobacter (Infections and infestations) | 1 (1) | 1 (1)
Perineal abscess (Infections and infestations) | 0 (0) | 1 (1)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 26 (28) | 17 (20)
Pharyngitis bacterial (Infections and infestations) | 0 (0) | 1 (1)
Plasmodium falciparum infection (Infections and infestations) | 3 (3) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 2 (2)
Post procedural infection (Infections and infestations) | 0 (0) | 1 (1)
Post procedural sepsis (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 3 (3) | 1 (1)
Pulpitis dental (Infections and infestations) | 13 (16) | 11 (11)
Pustule (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 1 (1)
Pyometra (Infections and infestations) | 0 (0) | 1 (1)
Rash pustular (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 38 (43) | 26 (28)
Respiratory tract infection viral (Infections and infestations) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 27 (29) | 20 (22)
Rhinovirus infection (Infections and infestations) | 1 (1) | 1 (1)
Salmonellosis (Infections and infestations) | 0 (0) | 1 (1)
Salpingitis (Infections and infestations) | 1 (1) | 2 (2)
Schistosomiasis (Infections and infestations) | 0 (0) | 1 (1)
Secondary syphilis (Infections and infestations) | 1 (1) | 0 (0)
Sexually transmitted disease (Infections and infestations) | 35 (38) | 45 (48)
Sinusitis (Infections and infestations) | 15 (18) | 11 (13)
Sinusitis bacterial (Infections and infestations) | 2 (2) | 4 (4)
Skin bacterial infection (Infections and infestations) | 1 (1) | 0 (0)
Skin candida (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 2 (2) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 17 (18) | 26 (30)
Syphilis (Infections and infestations) | 30 (32) | 26 (27)
Syphilis genital (Infections and infestations) | 4 (4) | 3 (4)
Tinea capitis (Infections and infestations) | 2 (2) | 3 (3)
Tinea cruris (Infections and infestations) | 2 (2) | 0 (0)
Tinea faciei (Infections and infestations) | 0 (0) | 3 (4)
Tinea infection (Infections and infestations) | 4 (4) | 3 (3)
Tinea manuum (Infections and infestations) | 3 (3) | 0 (0)
Tinea pedis (Infections and infestations) | 7 (8) | 2 (3)
Tinea versicolour (Infections and infestations) | 25 (27) | 18 (20)
Tonsillitis (Infections and infestations) | 63 (71) | 47 (52)
Tonsillitis bacterial (Infections and infestations) | 4 (4) | 5 (5)
Tooth abscess (Infections and infestations) | 4 (4) | 4 (4)
Tooth infection (Infections and infestations) | 1 (1) | 3 (3)
Trichomoniasis (Infections and infestations) | 20 (23) | 11 (12)
Tuberculous pleurisy (Infections and infestations) | 0 (0) | 1 (1)
Tubo-ovarian abscess (Infections and infestations) | 1 (1) | 0 (0)
Typhoid fever (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 240 (381) | 274 (403)
Upper respiratory tract infection bacterial (Infections and infestations) | 11 (11) | 13 (14)
Urinary tract candidiasis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 219 (347) | 203 (316)
Urinary tract infection bacterial (Infections and infestations) | 11 (11) | 7 (7)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1) | 0 (0)
Urogenital trichomoniasis (Infections and infestations) | 15 (15) | 6 (8)
Vaginal abscess (Infections and infestations) | 0 (0) | 3 (3)
Vaginal infection (Infections and infestations) | 27 (31) | 25 (30)
Vaginitis chlamydial (Infections and infestations) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 3 (3)
Varicella zoster virus infection (Infections and infestations) | 2 (2) | 0 (0)
Viral infection (Infections and infestations) | 6 (6) | 2 (2)
Viral parotitis (Infections and infestations) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 5 (5)
Viral rhinitis (Infections and infestations) | 10 (10) | 13 (16)
Viral sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Viral tonsillitis (Infections and infestations) | 0 (0) | 3 (3)
Viral upper respiratory tract infection (Infections and infestations) | 34 (40) | 38 (43)
Vulvovaginal candidiasis (Infections and infestations) | 127 (153) | 150 (188)
Vulvovaginal mycotic infection (Infections and infestations) | 1 (1) | 2 (2)
Vulvovaginitis (Infections and infestations) | 12 (12) | 9 (9)
Vulvovaginitis trichomonal (Infections and infestations) | 124 (146) | 109 (125)
Wound infection (Infections and infestations) | 0 (0) | 2 (2)
Wound sepsis (Infections and infestations) | 2 (2) | 3 (3)
Animal bite (Injury, poisoning and procedural complications) | 5 (5) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Any Event in SOC (Injury, poisoning and procedural complications) | 108 (129) | 122 (136)
Arthropod bite (Injury, poisoning and procedural complications) | 2 (2) | 5 (5)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 3 (3) | 6 (6)
Electrical burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Eye contusion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Eye injury (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Eyelid contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Face injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Human bite (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Iliotibial band syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inflammation of wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 4 (4) | 4 (4)
Ligament sprain (Injury, poisoning and procedural complications) | 3 (3) | 9 (9)
Limb injury (Injury, poisoning and procedural complications) | 9 (9) | 6 (6)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 14 (16) | 11 (11)
Periorbital haematoma (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Post procedural swelling (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Procedural pain (Injury, poisoning and procedural complications) | 14 (14) | 15 (15)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 11 (11) | 7 (7)
Skin wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 17 (17) | 27 (29)
Stab wound (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 6 (6) | 4 (4)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Traumatic arthritis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic ulcer (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 5 (5) | 1 (1)
Alanine aminotransferase increased (Investigations) | 51 (56) | 49 (57)
Amylase increased (Investigations) | 169 (217) | 149 (202)
Any Event in SOC (Investigations) | 1307 (4437) | 1331 (4502)
Aspartate aminotransferase increased (Investigations) | 40 (51) | 39 (44)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 1 (1)
Blood bicarbonate decreased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 12 (12) | 19 (25)
Blood calcium decreased (Investigations) | 5 (5) | 6 (7)
Blood calcium increased (Investigations) | 13 (13) | 5 (6)
Blood cholesterol increased (Investigations) | 4 (4) | 3 (3)
Blood creatine increased (Investigations) | 1 (1) | 5 (5)
Blood creatine phosphokinase increased (Investigations) | 85 (92) | 67 (72)
Blood creatinine decreased (Investigations) | 5 (5) | 2 (2)
Blood creatinine increased (Investigations) | 340 (610) | 330 (566)
Blood glucose decreased (Investigations) | 146 (180) | 146 (178)
Blood glucose increased (Investigations) | 75 (98) | 50 (66)
Blood phosphorus decreased (Investigations) | 58 (68) | 83 (104)
Blood phosphorus increased (Investigations) | 2 (2) | 0 (0)
Blood pressure diastolic increased (Investigations) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 14 (24) | 13 (14)
Blood pressure systolic increased (Investigations) | 1 (1) | 0 (0)
Blood triglycerides increased (Investigations) | 1 (1) | 3 (3)
Creatinine renal clearance decreased (Investigations) | 1166 (2812) | 1197 (2981)
Creatinine renal clearance increased (Investigations) | 0 (0) | 3 (3)
Gastric pH decreased (Investigations) | 2 (2) | 1 (1)
Glucose urine present (Investigations) | 0 (0) | 1 (1)
Haemoglobin decreased (Investigations) | 21 (24) | 20 (25)
Lipase increased (Investigations) | 52 (72) | 52 (68)
Low density lipoprotein increased (Investigations) | 12 (12) | 5 (5)
Lymphocyte count decreased (Investigations) | 9 (9) | 4 (7)
Neutrophil count decreased (Investigations) | 19 (22) | 20 (27)
Platelet count decreased (Investigations) | 16 (20) | 9 (11)
Protein urine present (Investigations) | 1 (1) | 0 (0)
Red blood cells urine positive (Investigations) | 2 (2) | 0 (0)
Urobilinogen urine increased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 8 (14) | 9 (11)
Weight increased (Investigations) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 3 (3) | 5 (5)
Abnormal loss of weight (Metabolism and nutrition disorders) | 85 (110) | 107 (167)
Abnormal weight gain (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Any Event in SOC (Metabolism and nutrition disorders) | 154 (200) | 194 (285)
Decreased appetite (Metabolism and nutrition disorders) | 34 (38) | 61 (67)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 4 (4)
Gout (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 11 (17) | 13 (13)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 15 (17) | 19 (22)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 6 (8)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Starvation (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Any Event in SOC (Musculoskeletal and connective tissue disorders) | 230 (335) | 220 (323)
Arthralgia (Musculoskeletal and connective tissue disorders) | 34 (37) | 39 (40)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 106 (130) | 112 (137)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 4 (4) | 7 (8)
Exostosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Extremity contracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 10 (10) | 9 (9)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 5 (5) | 5 (6)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 23 (27) | 21 (23)
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 43 (47) | 35 (43)
Myalgia (Musculoskeletal and connective tissue disorders) | 28 (32) | 21 (21)
Neck mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 5 (5)
Ochronosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 (22) | 16 (19)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Torticollis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Trismus (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertebral osteophyte (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 5 (5)
Any Event in SOC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 (8) | 8 (8)
Conjunctival neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Any Event in SOC (Nervous system disorders) | 309 (423) | 311 (467)
Cluster headache (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 10 (10) | 12 (13)
Dysgeusia (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 222 (283) | 222 (310)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 2 (2)
Migraine (Nervous system disorders) | 4 (4) | 4 (4)
Neuralgia (Nervous system disorders) | 2 (2) | 1 (1)
Neuritis (Nervous system disorders) | 1 (1) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 7 (7) | 8 (9)
Paraesthesia (Nervous system disorders) | 14 (16) | 21 (22)
Poor quality sleep (Nervous system disorders) | 1 (1) | 1 (1)
Post-traumatic headache (Nervous system disorders) | 1 (1) | 2 (2)
Psychogenic seizure (Nervous system disorders) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 4 (4) | 4 (4)
Sensory disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Sinus headache (Nervous system disorders) | 1 (1) | 1 (1)
Somnolence (Nervous system disorders) | 4 (5) | 4 (4)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Tension headache (Nervous system disorders) | 62 (82) | 70 (90)
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Any Event in SOC (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 3 (4)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Hyperemesis gravidarum (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
Morning sickness (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Retained products of conception (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Any Event in SOC (Product Issues) | 1 (1) | 0 (0)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Alcohol use disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Anger (Psychiatric disorders) | 0 (0) | 1 (2)
Anxiety (Psychiatric disorders) | 5 (5) | 4 (4)
Any Event in SOC (Psychiatric disorders) | 32 (39) | 31 (35)
Depression (Psychiatric disorders) | 3 (3) | 2 (2)
Depression suicidal (Psychiatric disorders) | 0 (0) | 1 (1)
Depressive symptom (Psychiatric disorders) | 0 (0) | 2 (2)
Emotional distress (Psychiatric disorders) | 6 (6) | 4 (4)
Generalised anxiety disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Grief reaction (Psychiatric disorders) | 1 (1) | 1 (1)
Insomnia (Psychiatric disorders) | 11 (12) | 12 (14)
Major depression (Psychiatric disorders) | 1 (1) | 2 (2)
Panic attack (Psychiatric disorders) | 1 (1) | 0 (0)
Panic disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Pica (Psychiatric disorders) | 1 (1) | 0 (0)
Post-traumatic stress disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (2) | 0 (0)
Stress (Psychiatric disorders) | 1 (1) | 1 (1)
Substance use disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0)
Any Event in SOC (Renal and urinary disorders) | 18 (19) | 20 (21)
Dysuria (Renal and urinary disorders) | 2 (2) | 3 (3)
Glycosuria (Renal and urinary disorders) | 2 (2) | 4 (5)
Haematuria (Renal and urinary disorders) | 2 (2) | 2 (2)
Polyuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 10 (10) | 11 (11)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Urine odour abnormal (Renal and urinary disorders) | 1 (1) | 0 (0)
Abnormal withdrawal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 3 (3) | 3 (3)
Any Event in SOC (Reproductive system and breast disorders) | 435 (734) | 419 (727)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 4 (4) | 5 (5)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical friability (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervical polyp (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cervix disorder (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Coital bleeding (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 150 (230) | 146 (212)
Dysmenorrhoea (Reproductive system and breast disorders) | 44 (51) | 61 (72)
Dyspareunia (Reproductive system and breast disorders) | 2 (2) | 2 (2)
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Endometriosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital rash (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Genital ulceration (Reproductive system and breast disorders) | 3 (3) | 5 (5)
Mammary duct ectasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 20 (27) | 18 (23)
Menorrhagia (Reproductive system and breast disorders) | 91 (110) | 91 (133)
Menstruation irregular (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Metrorrhagia (Reproductive system and breast disorders) | 92 (119) | 84 (110)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Nipple exudate bloody (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 12 (12) | 9 (10)
Polycystic ovaries (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Polymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premenstrual pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Premenstrual syndrome (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine cervical pain (Reproductive system and breast disorders) | 5 (5) | 7 (7)
Uterine spasm (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 83 (103) | 58 (90)
Vaginal haemorrhage (Reproductive system and breast disorders) | 14 (15) | 11 (11)
Vaginal ulceration (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Vulval ulceration (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 25 (32) | 22 (25)
Vulvovaginitis allergic (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Allergic pharyngitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Allergic sinusitis (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 11 (12)
Any Event in SOC (Respiratory, thoracic and mediastinal disorders) | 85 (97) | 77 (97)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 18 (19)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 13 (14)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (9)
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 17 (22)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (4)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Tonsillar inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 17 (19) | 14 (14)
Any Event in SOC (Skin and subcutaneous tissue disorders) | 187 (234) | 157 (207)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cold urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 25 (26) | 14 (15)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 34 (36) | 40 (47)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 9 (10) | 6 (7)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 5 (5)
Eczema (Skin and subcutaneous tissue disorders) | 7 (10) | 11 (12)
Hangnail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Intertrigo (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Lichen planus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Miliaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Perioral dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pityriasis rosea (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Prurigo (Skin and subcutaneous tissue disorders) | 11 (13) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 30 (36) | 28 (30)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 21 (23) | 20 (20)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash follicular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Rash papular (Skin and subcutaneous tissue disorders) | 10 (11) | 9 (9)
Rash pruritic (Skin and subcutaneous tissue disorders) | 8 (8) | 4 (4)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 17 (18) | 17 (17)
Any Event in SOC (Social circumstances) | 0 (0) | 3 (3)
Victim of crime (Social circumstances) | 0 (0) | 1 (1)
Victim of sexual abuse (Social circumstances) | 0 (0) | 2 (2)
Any Event in SOC (Vascular disorders) | 13 (13) | 22 (23)
Diastolic hypertension (Vascular disorders) | 1 (1) | 0 (0)
Essential hypertension (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 10 (10) | 20 (20)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT03164564/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/64/NCT03164564/SAP_001.pdf